CLINICAL TRIAL: NCT03997240
Title: A Randomized Wait-list Control Trial Evaluating the Effect of Team-based Applied Clinical Neuroscience Care on Self-reported Symptoms of Depression and Cerebellar Function in Adults With Medication-resistant Depression
Brief Title: Applied Clinical Neuroscience Care for Self-reported Symptoms of Depression and Cerebellar Function in Adults
Acronym: DEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Life University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: l-0012
Record Dates: First submitted 2019-06-24; First posted 2019-06-25 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-02

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Wait-list control (Other): Six-week wait list control
  Interventions: Procedure: Chiropractic Applied Clinical Neuroscience
- Immediate intervention (Experimental): Immediate treatment group
  Interventions: Procedure: Chiropractic Applied Clinical Neuroscience

INTERVENTIONS:
Procedure: Chiropractic Applied Clinical Neuroscience — Chiropractic Applied Clinical Neuroscience makes use of chiropractic care in addition to application of therapies designed to stimulate multisensory reintegration and cerebellar coordination. The multisensory reintegration and cerebellar therapies make use of the body's own sensory receptors as a target, with the purpose of realigning the brain's interpretation of different afferent signals. Observation of motor and autonomic output patterns during and after sensory stimulation afford the clinician real-time feedback, providing for adaptation of the sensory based protocol.

SUMMARY:
Pilot study design that operationalizes the multimodal manner of care while evaluating changes in depression symptoms, dysmetria, and balance for medication non-responders.

DETAILED DESCRIPTION:
Pilot study design that operationalizes the multimodal manner of care while evaluating changes in depression symptoms, dysmetria, and balance for medication non-responders. This research will provide an initial first step towards answering the following three research questions:

1. Does a multimodal chiropractic applied clinical neuroscience approach to care affect self-reported symptoms of depression?
2. Does a multimodal chiropractic applied clinical neuroscience approach to care affect dysmetria and balance control in a clinically depressed population?
3. Are changes in dysmetria and balance control correlated with a change in depressive symptoms.

ELIGIBILITY:
Inclusion Criteria:

* You are over the age of 18.
* You have been diagnosed with depression.
* You are currently taking medication for depression or have previously taken medication.
* You have been or were on your depression medication for at least 3 months.
* You feel/felt that the medication is/was not helping.

Exclusion Criteria:

* Had a lifetime history of severe neurologic or mental illness (e.g. schizophrenia or substance abuse)
* Are pregnant
* Have pending litigation or a recent history of spinal fracture, metastatic cancer, chiropractic care within the past month
* Present with contraindications to chiropractic care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2023-07-11 (Actual); Study Completion 2023-07-11 (Actual)

PRIMARY OUTCOMES:
P300 Auditory Evoked Potential task | 20 minutes
  Time-locked electroencephalography recording of the P300 event related potential. P300 testing involves placing electrodes on the participant's scalp while the individual is listening to a series to two different tones through headphones.

SECONDARY OUTCOMES:
Shift Balance Platform | 10 minutes
  Limits of stability test: For the limits of stability test the participant will be asked to lean forward, backward, left, and right. The participant will lean slowly in each direction at a self-determined speed and to a point where he or she feels is the maximum leaning distance without falling. The tests should take about 2 minutes but will vary based on the participant.

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Sullivan, DC, PhD, Principal Investigator — Life University
Locations (1):
- NeuroLife Institute, Marietta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No